CLINICAL TRIAL: NCT07041619
Title: Changes in Brain Activity as a Function of Scalp and Subcutaneous Electrical Stimulation Parameters in Epileptic Patients
Brief Title: Subcutaneous Intersectional Short Pulse Stimulation in Epileptic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Neunos ZRt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OGYÉI/9674/2021
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: Stimulation of pathological epileptiform brain activity (Experimental)
  Interventions: Device: Intersection short-pulse (ISP) stimulation

INTERVENTIONS:
Device: Intersection short-pulse (ISP) stimulation — The intervention aims to terminate pathological brain oscillations (i.e. epileptiform activity) in patients.

SUMMARY:
A subgaleal electrode-based system combined with the novel intersectional short-pulse (ISP) stimulation was developed to enable non-invasive, high-intensity neuromodulation. ISP consists of ultra-brief, distributed pulses to maximize electric field strength in target areas while minimizing adverse effects on non-target tissues. Early preclinical studies demonstrate its efficacy in disrupting pathological oscillations and reducing seizures in animal models. This study investigates how targeted electrical brain stimulation by ISP stimulation impacts brain activity in epilepsy patients. The research aims to determine if ISP stimulation delivered via electrodes placed outside and under the scalp can safely and effectively reduce seizure frequency and intensity. Participants include epilepsy patients who haven't responded adequately to medication and aren't eligible for surgery. By precisely tuning stimulation parameters and timing stimulation to specific seizure patterns detected by EEG monitoring, the study seeks to optimize this technique for therapeutic use. The goal is to establish safety and feasibility of this minimally invasive stimulation approach, as well as to achieve preliminary efficacy data thorugh the reduction of seizure durations.

DETAILED DESCRIPTION:
This clinical trial focuses on evaluating the safety, tolerability, and effectiveness of Intersectional Short Pulse (ISP) electrical stimulation in epilepsy patients. As a secondary outcome, the efficacy of ISP for reducing epileptic seizure duration and severity is also assessed. The ISP method utilizes electrodes implanted subcutaneously beneath the scalp, guided by MRI imaging for precise targeting.

The trial encompasses the following phases:

* Obtaining informed consents
* MRI scans are conducted to personalize electrode placement based on head anatomy.
* Electrodes are surgically implanted under general anesthesia.
* Following implantation, continuous EEG monitoring captures baseline seizure activity.
* Patients participate in stimulation tests to confirm tolerable ISP parameters.
* Patients participate in stimulation tests to confirm the feasibility of ISP stimulation triggered by epileptic seizures. An advanced seizure-detection algorithm (with close supervision) triggers stimulation to target seizures at their onset either, aiming to prevent their progression.
* Safety and tolerability are continuously assessed through clinical observations and participant feedback.
* Possible acute effects of ISP stimulation (i.e. reduction of seizure severity and duration or stopping seizures entirely) are also recorded as secondary outcomes.
* After concluding data recording, electrodes are explanted and the patients are emitted.
* Follow-up evaluations ensure long-term safety and monitor ongoing seizure activity post-treatment.
* Data processing: EEG data is rigorously analyzed, comparing seizure duration, severity and frequency before and after stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Patients with drug-resistant focal epilepsy who, after non-invasive or invasive EEG monitoring and neuropsychological, epilepsy protocol cranial MRI, or FDG-PET/CT or FDG-PET/MRI and/or ictal SPECT, have been declared unfit for resective epilepsy surgery by an interdisciplinary epilepsy team.
* Diagnosis of focal or idiopathic generalised epilepsy
* With antiepileptic drugs, 4 or more focal seizures per month, or frequent spike-wave activity on EEG - min 10 sec/hour.
* A patient who is fit to care for the wound and whose home environment this in terms of compliance and cleanliness

Exclusion Criteria:

* subjects under 18 years old
* If the patient is suitable for resective surgery or if there are questions about the patient's suitability for resective surgery of autoimmune aetiology
* Progressive brain lesions on MRI or a serious internal organ disease or coagulopathy considered serious by your doctor
* Subjects who have an electrical energy transmitting implant implanted in the brain or other organ(s), including pacemakers, intracardiac defibrillators and any device meeting this definition
* Pregnancy. Pregnancy should be checked by a pregnancy test for all women of childbearing potential
* Previous traumatic brain and skull injury, stroke are not exclusionary, but in all such cases the examining physician and the Neunos technical support team should be consulted
* The presence of metal implants is generally considered contraindicated. In all such cases, the investigating physician or the Neunos technical support team should be consulted

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Automatically Detected Seizures Successfully Treated with Closed-loop Subgaleal ISP Stimulation [Feasibility] | From enrollment to the end of treatment at maximum 12 weeks
  Intervention delivery rate (success rate of demonstrating the deliverability of the method as designed in the patient population, i.e. automatic seizure detection followed by ictal stimulation by subgaleal ISP stimulation)
Incidence and Severity of Treatment-Emergent Adverse Events of Subgaleal ISP stimulation [Safety] | From enrollment to the end of treatment at maximum 12 weeks
  Frequency (number) and severity (graded mild, moderate, severe) of all adverse events experienced by each patient during the treatment period.
Level of Subjective Discomfort associated with of subgaleal ISP stimulation [Tolerability] | From enrollment to the end of treatment at maximum 12 weeks
  Patient-reported subjective perception of stimulation intensity recorded on a Visual Analog Scale (VAS), ranging from 0 (no discomfort) to 10 (maximum discomfort). Higher scores indicate greater discomfort and worse tolerability.

SECONDARY OUTCOMES:
Efficacy of seizure termination by subgaleal ISP stimulation | From enrollment to the end of treatment at maximum 12 weeks
  Percent decrease in average seizure duration between stimulated (i.e. treated) and non-stimulated (i.e. control) seizures

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Neurosurgery and Neurointerventional Clinic, Budapest, Hungary

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT07041619/Prot_SAP_000.pdf